CLINICAL TRIAL: NCT01467154
Title: Does Ultra-High Dose i.v. N-acetylcysteine Prevent Contrast Nephropathy in Patients With Chronic Kidney Disease Undergoing Emergency Contrast Tomography.
Brief Title: Evaluation of Intravenous N-acetylcysteine to Prevent Contrast Media Induced Nephrotoxicity in an Emergency Center
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Poletti Pierre-Alexandre, MD, University Hospital, Geneva
Other Study IDs: 2008DR4057
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Nephrotoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group
- NAC group

SUMMARY:
The aim of the present study is to determine whether a high dose of intravenous NAC is efficient in preventing CN after emergency contrast injection in patients with renal failure.

DETAILED DESCRIPTION:
Prevention of acute kidney injury (AKI) post contrast injection remains mandatory given its association to morbidity and mortality1.

Contrast nephropathy (CN) was classically defined as an increase in 25% or more or absolute increase of 44 umol/l of creatinine levels within three days following contrast injection2. Markers such as cystatine C may be more sensitive to identify CN and also to correlate to mortality8 although a definition of CN using these markers is lacking.

In patients undergoing elective radiological procedures, CN can be prevented by hydration, withdrawal of diuretics and nephrotoxic drugs. N Acetylcysteine (NAC) has been proposed to protect against contrast nephropathy since 200013. While hydratation is clearly beneficial in preventing CIN14, the role of NAC administration is still uncertain and results of RCTs gave conflicting results regarding its effect15.

Intravenous N-acetylcysteine (NAC) may be the form of choice in emergency procedures given its rapid disponibility and its ease of administration in patients whose consciousness is altered or who can not eat.

The aim of the present study is therefore to determine whether 6000 mg of intravenous NAC is efficient in preventing CN after emergency contrast injection in CKD patients.

Inclusion criteria:

One hundred and thirty consecutive patients with an estimated GFR < 60 mL/min and an indication to undergo an emergent contrast-enhanced CT will be included in the study. Exclusion criteria: asthma, pregnancy, obstructive nephropathy and patient or family's refusal.

Patients will be blindly randomized by computer to either placebo (0.45% saline) or high dose (6000 mg) iv n-acétylcystéine (flumicil) iv diluted in 0.45% saline. All patients will receive intravenous hydration (250 ml NaCl 0.45% at least) before the CT scan and 1000 ml after the examination depending on clinical possibilities.

Creatinine and cystatine C serum levels will be collected one hour before CT scan and at day 2, 4 and 10. The T0 value will be the value measured before the CT-scan and not the baseline admission value in order to correct for differential hydratation due to different waiting time and hydratation before tomography. Serum Creatinine and Cystatine C will be measured by the Jaffe method, and by a nephelometric assay respectively.

Outcome measures:

The primary endpoint of the study will be the occurrence of contrast nephropathy at day 2, 4 or 10, defined as an increase of at least 25% and/or 44 umol/l in serum creatinine level or cystatine C levels at day 2, 4 or 10 compared to day 0. We will also assess the proportion of patients with contrast nephropathy regarding the biomarker used and according to AKIN criteria as well. D The AKIN criteria defined a stage 1 AKI as an increase in creatinine between 150% and 199% from baseline or an absolute increase of at least 26.2 umol/l, a stage 2 AKI as an increase between 200% and 299% from baseline and a stage 3 AKI as an increase of at least 300% from baseline or a creatinine concentration higher than 354 umol/l with an acute rise of at least 44 umol/l or initiation of RRT.

Secondary endpoints will be the mean increases in creatinine and cystatin C concentrations in days 2, 4 and 10 and the maximum increase during the time periods from day 2 to day 10 (peak increase).

ELIGIBILITY:
Inclusion Criteria:

* Renal failure and need of contrast enhanced CT

Exclusion Criteria:

* Asthma
* Pregnancy
* Obstructive nephropathy
* Patient or family's refusal
* In all patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency center patients
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
occurrence of contrast nephropathy at day 2, 4 or 10, which was defined as an increase of at least 25% and/or 44 umol/l in serum creatinine level or cystatine C levels at day 2, 4 or 10 compared to day 0. | 10 days

SECONDARY OUTCOMES:
mean increases in creatinine and cystatin C concentrations on days 2, 4 and 10 and maximum increase during the time periods from day 2 to day 10 (peak increase). | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexandre Poletti, MD, Principal Investigator — University Hospital, Geneva

REFERENCES:
- [Derived] Poletti PA, Platon A, De Seigneux S, Dupuis-Lozeron E, Sarasin F, Becker CD, Perneger T, Saudan P, Martin PY. N-acetylcysteine does not prevent contrast nephropathy in patients with renal impairment undergoing emergency CT: a randomized study. BMC Nephrol. 2013 Jun 3;14:119. doi: 10.1186/1471-2369-14-119. PMID 23731573